CLINICAL TRIAL: NCT04179240
Title: Using a Cartoon Questionnaire to Improve Consent of Children: A Randomized Controlled Trial
Brief Title: Using a Cartoon Questionnaire to Improve Consent of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Sijia Gu, Clinical Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SCMCIRB-K2016069
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Child Development; Ethics, Narrative
Keywords: biospecific nonspecimen specimen; child and adolescent; cartoon; questionnaire; concent
MeSH Terms: conditions — Narration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- audio and animated cartoon questionnaire group (Experimental): After a brief introduction to our survey, participants(children) were asked to complete a questionnaire on a professional platform named 'Wen juan xing app'(www.wjx.cn) with audio and animated cartoon questionnaire. The animation was an 8-minute cartoon video divided into different parts according to different questions. The first part of the animation was the introduction of biospecific nonspecimen specimen and our survey, while the other parts showed the content of the questionnaire about donating biospecific nonspecimen specimen in a vivid way. The background music built a relaxed and pleasant atmosphere, and some cartoon pictures were made into question options to simplify the understanding and data analysis.
  Interventions: Other: audio and animated cartoon questionnaire
- text questionnaire group (No Intervention): After a brief introduction to our survey, participants(children) were asked to complete a questionnaire on a professional platform named 'Wen juan xing app'(www.wjx.cn) with text questionnaire.
- Parent group (Other): After a brief introduction to our survey, participants(parent) were asked to complete a questionnaire on a professional platform named 'Wen juan xing app'(www.wjx.cn) with text questionnaire.
  Interventions: Other: audio and animated cartoon questionnaire

INTERVENTIONS:
Other: audio and animated cartoon questionnaire — participants were asked to complete a questionnaire audio and animated cartoon on a platform
  Arms: Parent group; audio and animated cartoon questionnaire group

SUMMARY:
In this study, a prospective, multicenter, randomized, and controlled trial will be performed to evaluate the effectiveness of an audio and animated cartoon questionnaire (AACQ) at improving child understanding and enhancing a positive attitude to participate in biospecific nonspecimen specimen donation.

DETAILED DESCRIPTION:
In this study, we will evaluate the effectiveness of an audio and animated cartoon questionnaire (AACQ) at improving child understanding and enhancing a positive attitude to participate in biospecific nonspecimen specimen donation. A prospective, multicenter, randomized, and controlled trial will be performed at some hospitals in China. Three hundred children will be randomly asked to participate in our survey to investigate the participants' willingness and attitudes for donating biospecific nonspecimen specimen.The participants will be randomly allocated to the AACQ group and the text questionnaire (TQ) group. A separate knowledge test to assess the amount of knowledge acquired is included in the questionnaires. Additionally, participants' demographic data and basic information will be also collected. In our present study, we aim to test whether an audio and animated cartoon could help the child to understand the information about our research of biospecific nonspecimen specimen donation, reduce differences in their understanding, and use that information to make an appropriate decision for themselves. Meanwhile, we will exam factors that may influence a Chinese child's willingness to donate biospecific nonspecimen specimen before pediatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients without obvious communication difficulties in the pediatric surgery wards were invited to participate in this survey.

Exclusion Criteria:

* Patients with obvious communication difficulties

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
correction rates | 1 hour after completing the questionnaire
  A knowledge test to assess the acquired comprehension of biospecific nonspecimen specimens donated was given at the end of the questionnaire
attitudes toward biospecific nonspecimen specimens | 1 hour after completing the questionnaire
  children's attitudes toward whether they would like to donate a particular kind of biospecific nonspecimen specimens

CONTACTS AND LOCATIONS:
Overall Officials: Shijian Liu, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No